CLINICAL TRIAL: NCT01060293
Title: Comparison of High-dose Furosemide, Low-dose Furosemide, and the Combination of Low-dose Furosemide and Low-dose Dopamine in Patients With Acute Decompensated Heart Failure
Brief Title: Dopamine in Acute Decompensated Heart Failure II
Acronym: DAD-HF II
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Safety issues in the LDFD-group (higher heart rate with dopamine)
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Gregory Giamouzis, Assistant Professor of Cardiology, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3975
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Heart Failure; Dopamine; Furosemide; Worsening Renal Function; Hypokalemia; Outcomes; Prognosis
MeSH Terms: conditions — Heart Failure; Hypokalemia | interventions — Furosemide; Dopamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-dose furosemide (Active Comparator): High-dose furosemide (HDF): 20 mg/h continuous IV administration for 8 hours
  Interventions: Drug: High-dose furosemide
- Low-dose furosemide (Active Comparator): Low-dose furosemide (LDF): continuous IV administration of 5 mg/h furosemide
  Interventions: Drug: Low-dose furosemide
- Low-dose furosemide combined with low-dose dopamine (Active Comparator): Low-dose furosemide combined with low-dose dopamine (LDFD): continuous IV administration of 5 mg/h furosemide combined with 5 μg/kg/min dopamine for a total of 8 hours
  Interventions: Drug: Low-dose furosemide combined with low-dose dopamine

INTERVENTIONS:
Drug: High-dose furosemide — High-dose furosemide (HDF): 20 mg/h continuous IV administration for 8 hours
  Arms: High-dose furosemide
Drug: Low-dose furosemide — Low-dose furosemide (LDF): continuous IV administration of 5 mg/h furosemide
  Arms: Low-dose furosemide
Drug: Low-dose furosemide combined with low-dose dopamine — Low-dose furosemide combined with low-dose dopamine (LDFD): continuous IV administration of 5 mg/h furosemide combined with 5 μg/kg/min dopamine for a total of 8 hours
  Arms: Low-dose furosemide combined with low-dose dopamine

SUMMARY:
The aim of this study is to compare the effects of 1) high-dose furosemide, 2) low-dose furosemide, and 3) low-dose furosemide combined with low-dose dopamine on diuresis, clinical status, renal function, electrolyte balance, length of stay, and 60-day post-discharge outcomes in patients hospitalized with acute decompensated heart failure.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of:

1. high-dose furosemide (HDF, 40 mg furosemide bolus IV, followed by continuous IV infusion of 20 mg/h for a total of 8 hours),
2. low-dose furosemide (LDF, 40 mg furosemide bolus IV, followed by continuous IV infusion of 5 mg/h furosemide for a total of 8 hours), and
3. low-dose furosemide combined with low-dose dopamine (LDFD, 40 mg furosemide bolus IV, followed by continuous IV infusion of 5 mg/h furosemide plus 5μg/kg/min dopamine for a total of 8 hours) on diuresis, perceived dyspnea, renal function, electrolyte balance, total length of stay, and 60-day post-discharge outcomes in patients hospitalized with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* patients with New York Heart Association (NYHA) functional class IV heart failure according to the American Heart Association (AHA) classification, namely dyspnea on minimal exertion or rest dyspnea, orthopnea, and paroxysmal nocturnal dyspnea,
* signs of congestion (third heart sound or pulmonary rales on physical examination),
* pulmonary congestion on chest x-ray,
* serum B-type natriuretic peptide levels > 400 pg/ml or NT-proBNP > 1500 pg/ml,
* echocardiographic documentation of systolic or diastolic dysfunction,
* age >18 years old,
* on medical therapy with an ACE-inhibitor and/or a β-blocker,
* experiencing an acute decompensation of known chronic HF,
* baseline oxygen saturation <90% on admission arterial blood gas

Exclusion Criteria:

* acute de novo HF;
* severe renal failure (serum creatinine >200 μmol/L or GFR <30 ml/min/1.73m2)
* admission systolic blood pressure <90 mm Hg;
* severe valvular disease;
* known adverse reactions to furosemide or dopamine;
* HF secondary to congenital heart disease;
* a scheduled procedure with a need for IV contrast dye;
* a scheduled cardiac surgery within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
1-year mortality or rehospitalization (all-cause, cardiovascular, non-cardiovascular, and due to worsening heart failure). | 1-year

SECONDARY OUTCOMES:
60-day mortality or rehospitalization (all-cause, cardiovascular, non-cardiovascular, and due to worsening heart failure). | 60-day post discharge
Novel indices of acute renal ischemia/injury (cystatin-C, KIM-1, NGAL) | Throughout hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Giamouzis, MD, Study Chair — Department of Cardiology, Larissa University Hospital, Larissa, Greece; Filippos Triposkiadis, MD, Study Chair — Department of Cardiology, Larissa University Hospital, Larissa, Greece
Locations (6):
- United States (2):
  - Division of Cardiology, Emory University Hospital, Atlanta, Georgia
  - The Cleveland Clinic Foundation, Cleveland, Ohio
- Greece (4):
  - First Department of Cardiology, University of Athens, Athens, Attica
  - Department of Cardiology, Larissa University Hospital, Larissa, Larissa
  - Department of Cardiology, Volos General Hospital, Volos, Magnesia
  - AHEPA University Hospital, Thessaloniki, Thessaloniki

REFERENCES:
- [Derived] Triposkiadis FK, Butler J, Karayannis G, Starling RC, Filippatos G, Wolski K, Parissis J, Parisis C, Rovithis D, Koutrakis K, Skoularigis J, Antoniou CK, Chrysohoou C, Pitsavos C, Stefanadis C, Nastas J, Tsaknakis T, Mantziari L, Giannakoulas G, Karvounis H, Kalogeropoulos AP, Giamouzis G. Efficacy and safety of high dose versus low dose furosemide with or without dopamine infusion: the Dopamine in Acute Decompensated Heart Failure II (DAD-HF II) trial. Int J Cardiol. 2014 Mar 1;172(1):115-21. doi: 10.1016/j.ijcard.2013.12.276. Epub 2014 Jan 10. PMID 24485633